CLINICAL TRIAL: NCT03487120
Title: Open Facet Joint Denervation in the Treatment of Low Back Pain -A Randomized Control Trial.
Brief Title: Open Facet Joint Denervation in the Treatment of Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. David Yen, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCTO
Record Dates: First submitted 2018-03-23; First posted 2018-04-03 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lumbar laminectomy (No Intervention)
- lumbar laminectomy with denervation of the facet joint (Active Comparator)
  Interventions: Procedure: facet joint denervation

INTERVENTIONS:
Procedure: facet joint denervation — Bipolar electrocautery
  Arms: lumbar laminectomy with denervation of the facet joint

SUMMARY:
A single blinded RCT for adult patients with spine pain. One group had a lumbar laminectomy with denervation of the facet joint at the level decompressed. The other group had a lumbar laminectomy without facet joint denervation. Both groups had their back pain and functional limitations measured using a 10 cm visual analogue scale and the Oswestry disability index (ODI). All measures were taken before surgery and at patients' 6, 12 and 24 week follow-up clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* aged 19 or older
* a diagnosis of spinal stenosis
* having neurogenic claudication
* complained of back pain for at least 3 months

Exclusion Criteria:

* previous surgery on their spine,
* fracture, systemic inflammatory disease,
* malignancies or an infection affecting their spine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Visual analog scale for pain (VAS) | change from baseline score at 24 weeks
  10 centimeter scale with a minimum of 0 indicating no pain and a maximum of 10 indicating worst pain.

SECONDARY OUTCOMES:
Change in Modified Oswestry Disability score (ODI) | change from baseline score at 24 weeks
  The ODI is divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale. The range of scores is 0 to a maximum of 60. The total score is multiplied by 2 and expressed as a percentage. A score of 0 to 20 points indicates minimal disability; 20 to 40 points, moderate disability; and 40 to 60 points, severe disability.

IPD SHARING:
Plan to Share IPD: No